CLINICAL TRIAL: NCT07322744
Title: Association Between Preoperative Lymphocyte-to-Monocyte Ratio and Postoperative Delirium According to Frailty Status in Older Surgical Patients: A Prospective Cohort Study
Brief Title: Preoperative Lymphocyte-to-Monocyte Ratio and Postoperative Delirium by Frailty Status in Older Surgical Patients
Status: Completed | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Yanhong Liu, Deputy Chief of administration, Anesthesiology, Chinese PLA General Hospital
Other Study IDs: LMR - POD
Record Dates: First submitted 2025-12-23; First posted 2026-01-07 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-11

CONDITIONS: Postoperative Delirium (POD); Frailty at Older Adults; Lymphocyte
Keywords: postoperative delirium; frailty; older surgical patients; lymphocyte-to-monocyte ratio
MeSH Terms: conditions — Emergence Delirium; Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- A retrospective cohort study based on prospectively collected data.: Patients were grouped according to the preoperative lymphocyte-to-monocyte ratio (LMR), calculated as the lymphocyte count divided by the monocyte count. Lymphocyte and monocyte values were obtained from the most recent preoperative laboratory test. Frailty was assessed one day before surgery using the FRAIL scale, which comprises five domains: fatigue, resistance, ambulation, illnesses, and weight loss. Each item is scored as 0 or 1, yielding a total score ranging from 0 to 5, with higher scores indicating greater frailty. Based on the total score, patients were categorized as robust (0 points), pre-frail (1-2 points), or frail (3-5 points).

SUMMARY:
Both frailty and a reduced preoperative lymphocyte-to-monocyte ratio (LMR) are known risk factors for postoperative delirium (POD). However, whether the relationship between LMR and POD varies by frailty status remains unclear. This study aimed to evaluate the frailty-stratified association between preoperative LMR and POD in older surgical patients.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥65 years;
* Underwent elective noncardiac, nonneurosurgical procedures;
* Completed the preoperative health and functional status questionnaire.

Exclusion Criteria:

* Severe dementia, language disorders, significant hearing or visual impairments, or coma;
* Cognitive function below the Mini-Mental State Examination thresholds (<18 for illiterate individuals, <21 for individuals with primary education, and <25 for individuals with secondary education or higher);
* Surgery performed under local anesthesia or monitored anesthesia care;
* Missing lymphocyte or monocyte count data;
* Missing postoperative delirium assessment;
* Incomplete preoperative FRAIL scale evaluation;
* Missing data for more than 20% of covariates.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients were grouped according to the preoperative lymphocyte-to-monocyte ratio (LMR) and were further stratified into subgroups based on frailty status, which was assessed one day before surgery using the FRAIL scale. Postoperative delirium was assessed using the 3-Minute Diagnostic Interview for Confusion Assessment Method (3D-CAM) for seven consecutive postoperative days or until hospital discharge, whichever occurred first.
Sampling Method: Non-Probability Sample
Enrollment: 6475 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
The primary outcome was the occurrence of postoperative delirium (POD). | POD assessment was performed twice daily for up to seven consecutive postoperative days or until hospital discharge, whichever occurred first.
  The primary outcome was the occurrence of POD, evaluated by trained researchers using the 3-Minute Diagnostic Interview for Confusion Assessment Method (3D-CAM).

CONTACTS AND LOCATIONS:
Locations (1):
- 28 Fuxing Road, Haidian District, Beijing, China

IPD SHARING:
Plan to Share IPD: No